CLINICAL TRIAL: NCT01496950
Title: Double-blind Randomized Clinical Trial to Evaluate Safety and Efficacy of Repetitive Transcranial Magnetic Stimulation in the Preventive Treatment of Chronic Migraine
Brief Title: Double-blind Randomized Clinical Trial of Transcranial Magnetic Stimulation in Chronic Migraine
Acronym: TMS-CHROMIG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Adriana Conforto, Professor of Neurology, MD PhD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIEP394-07
Record Dates: First submitted 2011-05-25; First posted 2011-12-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Chronic Migraine
Keywords: migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator: Active rTMS (Active Comparator): 10Hz active rTMS delivered to the left dorsolateral prefrontal cortex
  Interventions: Device: 10Hz active rTMS
- Placebo (Placebo Comparator): 10Hz placebo rTMS delivered to the vertex
  Interventions: Device: Placebo

INTERVENTIONS:
Device: 10Hz active rTMS — 10Hz active rTMS delivered to the left dorsolateral prefrontal cortex
  Other Names: Repetitive transcranial magnetic stimulation
  Arms: Active Comparator: Active rTMS
Device: Placebo — 10Hz placebo rTMS delivered to the vertex
  Other Names: Repetitive transcranial magnetic stimulation
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether active repetitive transcranial magnetic stimulation of the left dorsolateral prefrontal cortex is safe and effective for preventive treatment of chronic migraine, compared to placebo repetitive transcranial magnetic stimulation.

DETAILED DESCRIPTION:
Patients with chronic migraine according to the criteria of the International Headache Society will be randomized to either active repetitive transcranial magnetic stimulation of the left dorsolateral prefrontal cortex or placebo repetitive transcranial magnetic stimulation, in a total of 23 sessions of treatment (15 sessions in the first month and 8 sessions in the second month of treatment). Outcomes will be evaluated at baseline, after one, two months after treatment, and one month after end of treatment

ELIGIBILITY:
Inclusion Criteria:

* chronic migraine according to the criteria of the International Headache Society
* no change in prophylactic medication in the past 3 months

Exclusion Criteria:

* other neurological disorders
* bipolar disorder
* alcohol or drug dependence in the past 2 months
* suicidal ideation, psychotic symptoms
* contraindications to transcranial magnetic stimulation (cardiac pacemaker, implanted electronic devices, metal in the skull, skull fractures, history of seizures)
* use of antidepressants in the past 4 weeks
* pregnancy or lack of birth-control method in women of childbearing age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
number of days with pain per month | After all treatment sessions (total, 23 sessions within 60 days)

SECONDARY OUTCOMES:
adverse effects | After all treatment sessions (total, 23 sessions within 60 days)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Conforto, MD,PHD, Principal Investigator — Instituto Israelita de Ensino e Pesquisa Albert Einstein
Locations (1):
- Instituto Israelita de Ensino e Pesquisa Albert Einstein, São Paulo, Brazil